CLINICAL TRIAL: NCT04496895
Title: The Evaluation of Orange Peel Fermentation on Body Fat Lowering Efficacy in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201912030RSA
Record Dates: First submitted 2020-07-26; First posted 2020-08-03 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Overweight; Fatty Liver Disease
MeSH Terms: conditions — Overweight; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): consume 1 sachet per day for 2 months
  Interventions: Dietary Supplement: Placebo
- orange peel fermentation (Experimental): consume 1 sachet per day for 2 months
  Interventions: Dietary Supplement: orange peel fermentation

INTERVENTIONS:
Dietary Supplement: Placebo — consume 1 sachet per day for 2 months
  Arms: Placebo
Dietary Supplement: orange peel fermentation — consume 1 sachet per day for 2 months
  Arms: orange peel fermentation

SUMMARY:
To assess whether orange peel fermentation has the effect of reducing body fat in adults

DETAILED DESCRIPTION:
This is a double-blind and randomized study. Subjects are informed to consume the samples every day for 2 months. The clinical diagnosis item of overweight or fatty liver is evaluated by the doctor. The questionnaires are collected at every visit of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 20 and 65 who are willing to sign the consent form of the subject.
2. For those with BMI ≥ 24 or fatty liver, male body fat ≥ 25%, female body fat ≥ 30%.
3. Those who are not pregnant and are willing to cooperate with contraception during the trial period.
4. No history of cardiovascular disease, history of organ transplantation, history of epilepsy or convulsions, liver and kidney disease, malignant tumor, endocrine disease, mental disease, alcohol or drug abuse, or other major organic diseases (according to medical history).

Exclusion Criteria:

1. Pregnant women, people with a history of cardiovascular disease, organ transplantation, epilepsy or convulsions, liver and kidney disease, malignant tumors, endocrine diseases, mental illness, alcohol or drug abuse, and other major organic diseases (according to medical history).
2. No person who has received major surgery or bariatric surgery (according to medical history).
3. I have used drugs that affect body fat, waist circumference or significantly increase weight, such as systemic corticosteroids, tricyclic antidepressants, atypical psychiatric drugs, and mood stability in the current or 3 months before participating in the screening Drugs (according to medical history).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-11-12 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of body fat mass | Weeks 0, 4 and 8
  The body fat mass (kg) was assessed by InBody770
The change of Triglyceride | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of Triglyceride
The change of Total cholestrol | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of Total cholestrol
The change of HDL-cholestrol | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of HDL-cholestrol
The change of LDL-cholestrol | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of LDL-cholestrol
The change of body mass index (BMI) | Weeks 0, 4 and 8
  BMI is a measurement of a person's leanness or corpulence based on their height and weight, and is intended to quantify tissue mass.The body mass index (BMI, kg/m^2) and body mass (kg) were assessed by InBody770.
The change of body fat percentage | Weeks 0, 4 and 8
  The body fat percentage (%) was assessed by InBody770.
The change of visceral fat | Weeks 0, 4 and 8
  The visceral fat (10 cm^2) was assessed by InBody770.
The change of fasting glycemia | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of fasting glycemia
The change of aspartate aminotransferase | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of aspartate aminotransferase
The change of alanine aminotransferase | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of alanine aminotransferase
The change of albumin | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of creatine
The change of creatine | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of creatine
The change of uric acid | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of uric acid
The change of white blood cell | Weeks 0, 4 and 8
  Venous blood was sampled to measure concentrations of white blood cell

CONTACTS AND LOCATIONS:
Overall Officials: LIOU JYH-MING, Doctor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan